CLINICAL TRIAL: NCT00002562
Title: EVALUATION OF PACLITAXEL (TAXOL) IN PERSISTENT OR RECURRENT NON-SQUAMOUS CELL CARCINOMA OF THE CERVIX AND VAGINA
Brief Title: Paclitaxel in Treating Patients With Advanced, Refractory, or Recurrent Cervical or Vaginal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000063506; GOG-128B
Record Dates: First submitted 1999-11-01; First posted 2004-08-10 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2005-12

CONDITIONS: Cervical Cancer; Vaginal Cancer
Keywords: recurrent cervical cancer; recurrent vaginal cancer; vaginal clear cell adenocarcinoma; cervical adenocarcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients with advanced, refractory, or recurrent cervical or vaginal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the frequency and duration of objective response, duration of progression-free interval, and survival of patients treated with paclitaxel for advanced, persistent, or recurrent clear cell adenocarcinoma of the vagina and cervix who have failed higher priority treatment protocols. II. Determine the frequency and severity of observed adverse effects on this study.

OUTLINE: Single-Agent Chemotherapy. Paclitaxel, TAX, NSC-673089.

PROJECTED ACCRUAL: 25 evaluable patients per histologic stratum will be accrued over 10-12 months for the nonsquamous cell carcinoma stratum and over 23 months for the clear cell adenocarcinoma stratum. If more than 3 patients in a given stratum respond, an additional 25 patients will be accrued to that stratum. As of 07/95, the study is open only to patients with clear cell adenocarcinoma of the vagina or cervix.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced, persistent, or recurrent clear cell adenocarcinoma of the vagina or cervix Documented disease progression after local therapy required Disease must be considered incurable Bidimensionally measurable disease required by physical examination or medical imaging

PATIENT CHARACTERISTICS: Age: Any age Performance status: GOG 0-2 Hematopoietic: WBC at least 3,000 AGC at least 1,500 Platelets at least 100,000 Hepatic: Bilirubin no more than 1.5 times normal AST no more than 3 times normal Alkaline phosphatase no more than 3 times normal Renal: Creatinine no more than 2.0 mg/dL Other: Not eligible for a higher priority GOG protocol No significant infection No prior or concomitant second malignancy except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: At least 3 weeks since therapy directed at malignancy Biologic therapy: Not specified Chemotherapy: No more than 1 prior chemotherapy regimen (either single or combination cytotoxic drug therapy) No prior paclitaxel Recovery from prior chemotherapy required Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy for recurrent disease except a low dose, single fraction used to abrogate menorrhagia Recovery from prior radiotherapy required Surgery: Recovery from prior surgery required

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1994-03; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Curtin, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (50):
- United States (50):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Women's Cancer Center, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Result] Curtin JP, Blessing JA, Webster KD, Rose PG, Mayer AR, Fowler WC Jr, Malfetano JH, Alvarez RD. Paclitaxel, an active agent in nonsquamous carcinomas of the uterine cervix: a Gynecologic Oncology Group Study. J Clin Oncol. 2001 Mar 1;19(5):1275-8. doi: 10.1200/JCO.2001.19.5.1275. PMID 11230468